CLINICAL TRIAL: NCT00003255
Title: Phase II Study of Continuous Infusion Carboplatin and Topotecan in the Treamtment of Relapsed Acute Myelogenous Leukemia (AML)
Brief Title: Carboplatin Plus Topotecan in Treating Patients With Relapsed Acute Myelogenous Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-968151; CDR0000066143 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-11-01; First posted 2004-05-20 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: Leukemia
Keywords: recurrent adult acute myeloid leukemia; secondary acute myeloid leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute | interventions — Carboplatin; Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- topotecan + carboplatin (Experimental): Patients receive continuous intravenous infusions of topotecan and carboplatin for 5 days. Treatment repeats every 3-4 weeks during induction (two courses) and every 6-10 weeks during consolidation. No more than four courses of treatment are given. Patients are followed every 6 months for 5 years.
  Interventions: Drug: carboplatin; Drug: topotecan hydrochloride

INTERVENTIONS:
Drug: carboplatin
Drug: topotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining carboplatin and topotecan in treating patients with relapsed acute myelogenous leukemia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the efficacy of a 5-day continuous infusion of carboplatin and topotecan in patients with relapsed and refractory acute myelogenous leukemia (AML). II. Assess the toxic effects of this treatment in these patients.

OUTLINE: Patients receive continuous intravenous infusions of topotecan and carboplatin for 5 days. Treatment repeats every 3-4 weeks during induction (two courses) and every 6-10 weeks during consolidation. No more than four courses of treatment are given. Patients are followed every 6 months for 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Previously established diagnosis of acute myelogenous leukemia: Failure to achieve a complete remission with initial induction regimen First relapse within 1 year of initial complete remission Failure to achieve complete remission with one or two courses of reinduction therapy at first relapse Second relapse after no more than two different induction regimens Chemotherapy-related leukemia with unfavorable cytogenetics No active CNS leukemia Not eligible for allogeneic bone marrow transplant from related donor

PATIENT CHARACTERISTICS: Age: 18 to 74 Performance status: ECOG 0-2 Life expectancy: At least 4 weeks Hematopoietic: Not specified Hepatic: Bilirubin no greater than upper limit of normal (ULN) (unless elevation due to AML) Renal: Creatinine no greater than 0.3 mg/dL above ULN Cardiovascular: No myocardial infarction within the past 3 months No congestive heart failure No poorly controlled cardiac arrhythmia Other: Not pregnant or nursing Fertile patients must use adequate contraception No psychosis No active systemic infections

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Recovered from the toxic effects of previous chemotherapy At least 3 days since hydroxyurea Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: Not specified Other: No prior or concurrent aminoglycosides or amphotericin B within past 7 days

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 1999-11; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
overall survival | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Scott H. Kaufmann, MD, PhD, Study Chair — Mayo Clinic